CLINICAL TRIAL: NCT04094103
Title: Integrated Cardiovascular and Metabolic Effects of Strawberry Consumption in Overweight and Obese Individuals
Brief Title: Strawberry Consumption in Overweight and Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Ade, M.S., Ph.D. (Other)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor-Investigator, Carl Ade, M.S., Ph.D., Co-Principal Investigator, Kansas State University
Organization: Kansas State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Pro9736
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The supplement and placebo will be distributed to the individual by a member of the research team who is not involved with data collection or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active strawberry powder (Experimental): Participants will consume a 39g freeze-dried active strawberry powder beverage once per day for 4-weeks.
  Interventions: Dietary Supplement: Active strawberry powder
- Placebo strawberry powder (Placebo Comparator): Participants will consume a 39g freeze-dried strawberry powder placebo beverage once per day for 4-weeks.
  Interventions: Dietary Supplement: Placebo strawberry powder
- Mixed active/placebo strawberry powder (Active Comparator): Participants will consume a 39g mixed active/placebo strawberry powder beverage once per day for 4-weeks.
  Interventions: Dietary Supplement: Mixed strawberry powder

INTERVENTIONS:
Dietary Supplement: Active strawberry powder — Participants will drink a strawberry beverage with active ingredients once a day during the 4-week intervention period.
  Arms: Active strawberry powder
Dietary Supplement: Placebo strawberry powder — Participants will drink a strawberry placebo beverage once a day during the 4-week intervention period.
  Arms: Placebo strawberry powder
Dietary Supplement: Mixed strawberry powder — Participants will drink a mixed strawberry beverage with active ingredients and placebo once a day during the 4-week intervention period.
  Arms: Mixed active/placebo strawberry powder

SUMMARY:
Our proposal represents an integrated approach to determining the cardiovascular and metabolic effects of strawberry consumption in adults who have high risk for cardiometabolic disease.

DETAILED DESCRIPTION:
The current proposal aims to fill some of these important research gaps with regard the dose and time-course of strawberry consumption in a population where dietary intervention may of particular benefit for both primary and secondary prevention of cardiovascular and metabolic disease. Participants will participate in a double blind, placebo-controlled, randomized crossover trial. Following a 10-day run-in where no berries are consumed, participants will be randomized via Latin-square design, to three different daily strawberry powder conditions for 4-weeks at a time, with a 7 day washout between conditions.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese by BMI (25.0-34.9kg/m2),
* Borderline-high LDL-cholesterol (130-159mg/dL),
* Normal or elevated blood pressure ((≤129mmHg/≤80mmHg)

Exclusion Criteria:

* known allergy or intolerance to strawberries
* taking any medications for chronic diseases including anti-inflammatory, anti-hypertensive, lipid-lowering, glucose-controlling, or steroidal medications
* taking any supplements that might affect outcomes of the study including anti-oxidant or fish-oil supplements
* having anemia or any liver, thyroid, renal conditions
* current smoker or user of tobacco products, or use within the past three months
* consuming alcohol (>1-2 drinks/day) on a regular basis
* currently pregnant or lactating
* having elevated blood pressure ≥130mmHg/≥80mmHg
* presence of diagnosed diabetes mellitus, inflammatory disease, atherosclerotic disease, or other relevant chronic conditions
* total cholesterol ≥240mg/dL
* hemoglobin normal range values for males (between 13.0-17.5g/dL) and females (between 12.5-15.5g/dL)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipids | Week 0, 4, 5, 9, 10, and 14
  Total cholesterol (TC), LDL-c , VLDL-c, HDL-c , triglycerides (TG) from blood sample in a fasted state and following consumption of a meal

SECONDARY OUTCOMES:
Change in glucose and insulin response | Week 0, 4, 5, 9, 10, and 14
  Glucose, insulin, and c-peptide obtained from blood sample in a fasted state and in response to a meal
Change in oxidixed LDL | Week 0, 4, 5, 9, 10, and 14
  Obtained from blood sample in a fasted state and following consumption of a meal
Change in homeostatic model assessment for insulin resistance | Week 0, 4, 5, 9, 10, and 14
  Calculated from fasting glucose and insulin values
Change in inflammation | Week 0, 4, 5, 9, 10, and 14
  hs-CRP and IL-6 will be assessed in the fasted state from plasma
Change in arterial stiffness | Week 0, 4, 5, 9, 10, and 14
  Determined via changes in carotid artery stiffness calculated from simultaneous measurements of carotid artery diameter and pressure-waveforms
Change in blood pressure (resting and 24-hr) | Week 0, 4, 5, 9, 10, and 14
  Evaluated via automated sphygmomanometer. 24-hr ambulatory blood pressure is taken at 20-30 minute intervals over a 24hr period while the individual goes about their normal activities and while sleeping.
Change in endothelial function | Week 0, 4, 5, 9, 10, and 14
  Flow mediated dilation (FMD) assessed via a non-invasive 2D Doppler ultrasound following a 5-min period of arterial occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rosenkranz, PhD, Principal Investigator — Kansas State University
Locations (1):
- Lafene Health Center, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No